CLINICAL TRIAL: NCT03833063
Title: Glabellar Botulinum Toxin Injections for the Treatment of Geriatric Depression
Acronym: BOTDEP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: recruitment difficulties due to COVID19
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019BR
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder; Major Depressive Episode; Treatment Resistant Depression
Keywords: botulinumtoxin; botox; depression; geriatric depression; depression in older adults; depression in the elderly; old age depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: placebo controlled, randomized, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): injections with sodium chloride
  Interventions: Drug: Placebos
- botulinum toxin A (Active Comparator): injections with botulinum toxin A
  Interventions: Drug: botulinum toxin A

INTERVENTIONS:
Drug: botulinum toxin A — glabellar injections with botulinum toxin A
  Arms: botulinum toxin A
Drug: Placebos — glabellar injections with sodium chloride
  Other Names: sodium chloride
  Arms: placebo

SUMMARY:
The effectiveness of glabellar injection of botulinum toxin type A (BTA) in treating depression has not yet been investigated in elderly patients. The study aims in addressing the question if glabellar injection of BTA is effective in treating geriatric depression.

DETAILED DESCRIPTION:
Feedback from facial expressions is known to influence emotional experience. Treatment of muscles involved in facial expression of sadness, anger or anxiety with botulinumtoxin showed a quick, strong and sustained improvement in the symptoms of depression. As considerable proportion of patients do not sufficiently respond to existing treatment options. Especially in the elderly current treatments show limited response or are associated with side effects. Injections with BTA are considered as a very safe treatment without lasting side effects. The aim of the study is to investigate effectiveness of BTA in treating major depression in the elderly in a cross-over designed, placebo-controlled manner.

ELIGIBILITY:
Inclusion criteria: Clinically relevant depressive symptoms ( defined as MADRS > 12)

Exclusion criteria: cognitive deficits that impair the participant´s ability to provide written informed consent severe depression MADRS >34 suicidality treatment with more than 3 psychotropic medications recent changes (4 weeks) in current psychotropic medication previous treatment with study drug active substance abuse bipolar disorder schizophrenia unstable medical condition usage of warfarin or NOAC bleeding disorder known hypersensitivity to study drog or any of the excipients of the formulation myasthenia gravis or Eaton Lambert syndrome presence of infection at the proposed injection sites

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Severity og depressive symptoms, response to treatment | 16 weeks
  Response to treatment, as defined as a 50% or greater decrease in Montgomery Aasberg Depression Rating Scale (MADRS) from baseline
  Montgomery-Åsberg Depression Rating Scale The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire to measure the severity of depressive episodes in patients with mood disorders.
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.[4] The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
  Usual cutoff points are:
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.

SECONDARY OUTCOMES:
remission | 16 weeks
  remission rate, as defined by a Montgomery Aasberg Depression Rating Scale MADRS score of 10 or lower
severity of depressive symptoms, self-rated Geriatric Depression Scale (GDS) | 16 weeks
  severity of depressive symptoms, self-rated Geriatric Depression Scale (GDS) In the Geriatric Depression Scale, questions are answered "yes" or "no." A five-category response set is not utilized in order to ensure that the scale is simple enough to be used when testing ill or moderately cognitively impaired individuals, for whom a more complex set of answers may be confusing, or lead to inaccurate recording of responses.
  The scale consists of 30 yes/no questions. Each question is scored as either 0 or 1 points. The following general cutoff may be used to qualify the severity:
  normal 0-9, mild depressives 10-19, severe depressives 20-30.
quality of life, as assessed with QOL-AD | 16 weeks
  quality of life, as assessed with the questionnaire QOL-AD Use of the QOL-AD for measuring quality of life in people with dementia Scoring instructions for QOL-AD: Points are assigned to each item as follows:poor=1,fair=2,good=3,excellent=4. The total score is the sum of all 13 items.
safety/tolerability | 16 weeks
  Incidence of Treatment-Emergent Adverse Events, as assessed by number in registration of AE/SAE

IPD SHARING:
Plan to Share IPD: No